CLINICAL TRIAL: NCT00389506
Title: A Pilot Study of Anti-Tac(Fv)-PE38 (LMB-2) Immunotoxin for Treatment of CD25 Positive Hodgkin's Disease After Fludarabine and Cyclophosphamide
Brief Title: Fludarabine and Cyclophosphamide Followed By LMB-2 Immunotoxin in Treating Patients With Hodgkin's Lymphoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: 060240; 06-C-0240; NCI-P6761; NCI-7835; CDR0000508789
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Lymphoma
Keywords: stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — B3(Fv)-PE38KDEL recombinant immunotoxin; Cyclophosphamide; fludarabine phosphate

INTERVENTIONS:
Biological: LMB-2 immunotoxin
Drug: cyclophosphamide
Drug: fludarabine phosphate
Other: pharmacological study

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. LMB-2 immunotoxin can find cancer cells and kill them without harming normal cells. Giving fludarabine and cyclophosphamide followed by LMB-2 immunotoxin may kill more cancer cells.

PURPOSE: This clinical trial is studying how well giving fludarabine and cyclophosphamide followed by LMB-2 immunotoxin works in treating patients with Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of pretreatment with fludarabine phosphate and cyclophosphamide in preventing neutralization of antibodies in patients with CD25-positive Hodgkin's lymphoma.

Secondary

* Determine the response rate in patients treated with LMB-2 immunotoxin.
* Determine the response duration in patients receiving this treatment.
* Correlate serum levels of LMB-2 immunotoxin with toxicity and response in these patients.
* Assess the development of neutralizing antibodies and the effect of these antibodies on blood levels of LMB-2 immunotoxin and toxicity.
* Correlate soluble Tac-peptide levels with treatment response in these patients.

OUTLINE: This is a nonrandomized, pilot study.

Patients receive fludarabine phosphate IV over 30 minutes and cyclophosphamide IV over 60 minutes on days 1-4 and filgrastim (G-CSF) subcutaneously once daily beginning on day 5 and continuing until blood counts recover.

Beginning 4 weeks after completion of chemotherapy, patients receive LMB-2 immunotoxin IV over 30 minutes on days 1, 3, and 5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression.

Blood is obtained prior to and after chemotherapy and then periodically during LMB-2 immunotoxin therapy for pharmacokinetic studies to measure lymphocyte subsets.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histopathologically confirmed CD25+ Hodgkin's lymphoma

  * At least 20% of the malignant cells positive by immunohistochemistry
  * Stage II-IV disease
* Meets the following criteria:

  * Failed standard chemotherapy
  * Not eligible for curative salvage radiotherapy or chemotherapy
  * Not eligible for or refused bone marrow transplantation
* Measurable disease
* No patient whose serum neutralizes LMB-2 immunotoxin in tissue culture, due either to antitoxin or antimouse-IgG antibodies
* No patient whose serum neutralizes > 75% of the activity of 1 µg/mL of LMB-2 immunotoxin

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 50,000/mm³
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* ALT and AST ≤ 2.5 times upper limit of normal
* Albumin ≥ 3.0 g/dL
* Bilirubin ≤ 2.2 mg/dL (< 5 mg/dL if Gilbert's syndrome is present)
* Creatinine ≤ 1.4 mg/dL OR creatinine clearance ≥ 50 mL/min
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would limit study compliance
* No HIV or hepatitis C positivity

  * Hepatitis B surface antigen positivity allowed provided patient is receiving lamivudine
* LVEF ≥ 45%
* DLCO ≥ 50% of normal OR FEV_1 ≥ 60% of normal
* No active second malignancy requiring treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No systemic cytotoxic chemotherapy within the past 4 weeks
* No systemic steroids (except stable doses of prednisone ≤ 20 mg/day) within the past 4 weeks
* No monoclonal antibody therapy within the past 12 weeks
* No prior LMB-2 immunotoxin
* No concurrent warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-09; Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of using fludarabine phosphate and cyclophosphamide to decrease neutralizing antibodies

SECONDARY OUTCOMES:
Response rate
Response duration
Correlation of serum levels of LMB-2 immunotoxin with toxicity and response
Development of neutralizing antibodies and its effect on blood level of LMB-2 immunotoxin and toxicity
Correlation of soluble Tac-peptide with treatment response

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kreitman, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States